CLINICAL TRIAL: NCT04528199
Title: A Phase 1 Study of [18F]FLOR (FC303) PET/CT Imaging in Patients With Prostate Cancer
Brief Title: [18F]FLOR (FC303) PET/CT Imaging in Patients With Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Principal Investigator decided to terminate the study because the PI left Hopkins.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: FutureChem (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J19145; IRB00231620 (Other: JHM IRB)
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Prostate Cancer
Keywords: [18F]FLOR; PET/CT; prostate cancer; J19145
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]FLOR (FC303) (Experimental): [18F]FLOR (FC303) PET/CT imaging.
  Interventions: Drug: [18F]FLOR (FC303) Injection

INTERVENTIONS:
Drug: [18F]FLOR (FC303) Injection — Single dose of 10 ±1 millicurie (mCi) of [18F]FLOR (FC303) injection followed by the PET/CT scan.

SUMMARY:
The study is an open label, single-arm study designed to evaluate the safety and diagnostic performance of [18F]FLOR (FC303) PET/CT imaging to determine the presence or absence of metastatic prostate cancer. .

DETAILED DESCRIPTION:
This research is being done to determine whether the radioactive compound called [18F]FLOR (FC303) is safe and well-tolerated in patients with metastatic prostate cancer.

Participants in this study will have tests, exams and procedures that are for study purposes. Participants will be in this study up to one month which will include up to three clinic visits.

Eligible patients diagnosed with metastatic prostate cancer will undergo a [18F]FLOR (FC303) PET-CT scan. This is the imaging procedure to assess where [18F]FLOR (FC303) has accumulated in the body.

ELIGIBILITY:
Inclusion Criteria:

* Males ≥18 years of age.
* Subjects provide signed informed consent and confirm that they are able and willing to comply with all protocol requirements.
* Histologically confirmed adenocarcinoma of the prostate.
* Radiologic evidence of local recurrence or new or progressive metastatic disease demonstrated on anatomical imaging (CT, or MRI), or whole-body bone scan within 4 weeks of Day 1.
* At least 2 weeks must have elapsed between last anti-cancer treatment administration and the imaging day. Imaging day will be scheduled before initiation of new systemic therapy for recurrent and/or progressive metastatic disease
* Screening clinical laboratory values within normal limits or judged not clinically significant by the investigator.

Exclusion Criteria:

* Subjects administered any radioisotope within five physical half-lives prior to study drug injection.
* Subjects with any medical condition or other circumstances that, in the opinion of the investigator, compromise obtaining reliable data, achieving study objectives, or completion.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
Incidence of study drug emergent adverse events | Up to 10 days post-study drug dosing
  Incidence of study drug emergent adverse events will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Rowe, M.D., Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States